CLINICAL TRIAL: NCT01890252
Title: Prospective, Randomized Crossover Study Of The Hyper-CL™ Lens (Hyper Osmotic Contact Lens) In Subjects Suffering From Corneal Edema
Brief Title: Hyper-CL™ Lens (Hyper Osmotic Contact Lens) In Subjects Suffering From Corneal Edema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eye-yon Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ECL00005
Record Dates: First submitted 2013-06-25; First posted 2013-07-01 (Estimated); Last update posted 2021-11-11 (Actual); Status verified 2019-02

CONDITIONS: Corneal Edema
MeSH Terms: conditions — Corneal Edema | interventions — Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Hyper CL (Experimental): Hyper osmotic contact lens
  Interventions: Device: Hyper CL
- Hyper CL + Saline solution (Experimental): combined treatment of hyper osmotic contact lens+ hypertonic solution
  Interventions: Device: Hyper CL; Drug: saline solution
- saline solution (Active Comparator): hypertonic solution
  Interventions: Drug: saline solution

INTERVENTIONS:
Device: Hyper CL — The Hyper CL is hyper osmotic contact lens that absorb fluids from the cornea and by that reduces corneal edema.
  Arms: Hyper CL; Hyper CL + Saline solution
Drug: saline solution — saline solution of 5% NaCl
  Other Names: hyper-tonic solution
  Arms: Hyper CL + Saline solution; saline solution

SUMMARY:
The Hyper-CL™ lenses are indicated for therapeutic use as a bandage to protect the corneal surface and to relieve corneal pain in the treatment of acute or chronic ocular pathologies, such as bullous keratopathy, corneal erosions, entropion, corneal edema, and corneal dystrophies as well as post-surgical conditions resulting from cataract extraction and corneal surgery. The lenses may be prescribed for daily wear with removal for cleaning and disinfection (chemical, not heat) prior to reinsertion, as recommended by the eye care professional.

In addition Hyper-CL™ contact lenses can also provide optical correction during healing if required.

Prospective open-label, randomized, crossover clinical study To evaluate the safety and efficacy of the Hyper-CL™ lens in subjects suffering from corneal edema.

This study is designed to evaluate the efficacy of the Hyper-CL™ lens contact lens on corneal edema thickness as compared with salt solution treatment only in subjects suffering from corneal edema.

Treatment with the Hyper-CL™ lens may result with greater reduction in edema thickness as compared with treatment with salt solution only in subjects suffering from corneal edema.

Men and women suffering from a decrease in vision due to corneal edema that meet the inclusion/exclusion criteria and provide written Informed Consent will be enrolled in the study.

A total of 25 subjects will be enrolled. Each subject will be treated with:

* Treatment A: Hyper-CL™ lens only (7 days)
* Treatment B: Hyper-CL™ lens + salt solution (7 days)
* Treatment C: salt solution only (7 days) One week (7 days) of washout without any treatment will be between treatments. Subject will be equally allocated (with a 1:1:1:1:1:1 ratio) to one of the following 6 crossover regimen based on a randomization scheme with blocks stratified by center: C-A-B; B-C-A; A-B-C; C-B-A; B-A-C; A-C-B.

Up to 2 centers will participate in this study. Each subject will be followed from baseline to 42 days. All Subjects will come for a clinic visit at 7, 14, 21, 28, 35 and 42 days post first treatment.

Completion of active enrolment is anticipated to last approximately 6 months. The primary end point will be achieved when the final study subject has completed 42 day follow-up.

DETAILED DESCRIPTION:
Prospective, randomized crossover study of the Hyper-CL™ lens (Hyper osmotic Contact Lens) in subjects suffering from corneal edema Hyper-CL™ lens (Hyper osmotic Contact Lens) The Hyper-CL™ lenses are indicated for therapeutic use as a bandage to protect the corneal surface and to relieve corneal pain in the treatment of acute or chronic ocular pathologies, such as bullous keratopathy, corneal erosions, entropion, corneal edema, and corneal dystrophies as well as post-surgical conditions resulting from cataract extraction and corneal surgery. The lenses may be prescribed for daily wear with removal for cleaning and disinfection (chemical, not heat) prior to reinsertion, as recommended by the eye care professional.

In addition Hyper-CL™ contact lenses can also provide optical correction during healing if required.

Prospective open-label, randomized, crossover clinical study To evaluate the safety and efficacy of the Hyper-CL™ lens in subjects suffering from corneal edema.

This study is designed to evaluate the efficacy of the Hyper-CL™ lens contact lens on corneal edema thickness as compared with salt solution treatment only in subjects suffering from corneal edema.

Treatment with the Hyper-CL™ lens may result with greater reduction in edema thickness as compared with treatment with salt solution only in subjects suffering from corneal edema.

Men and women suffering from a decrease in vision due to corneal edema that meet the inclusion/exclusion criteria and provide written Informed Consent will be enrolled in the study.

A total of 25 subjects will be enrolled. Each subject will be treated with:

* Treatment A: Hyper-CL™ lens only (7 days)
* Treatment B: Hyper-CL™ lens + salt solution (7 days)
* Treatment C: salt solution only (7 days) One week (7 days) of washout without any treatment will be between treatments. Subject will be equally allocated (with a 1:1:1:1:1:1 ratio) to one of the following 6 crossover regimen based on a randomization scheme with blocks stratified by center: C-A-B; B-C-A; A-B-C; C-B-A; B-A-C; A-C-B.

Up to 2 centers will participate in this study. Each subject will be followed from baseline to 42 days. All Subjects will come for a clinic visit at 7, 14, 21, 28, 35 and 42 days post first treatment.

Completion of active enrolment is anticipated to last approximately 6 months. The primary end point will be achieved when the final study subject has completed 42 day follow-up.

The frequency and severity of all treatment-related adverse events, during and after using the Hyper-CL™ lens. Adverse events will be assessed on a continuous basis from the first procedure through the study completion at 42 days. Related adverse events include: infectious keratitis, allergic or toxic inflammatory reaction, significant increase in corneal edema.

Percent of subjects with corneal thickness decrease by at least 8% following treatment with the Hyper-CL™ lens + salt solution.

* Corneal thickness decrease following treatment with the Hyper-CL™ lens + salt solution
* Percent of subjects with corneal thickness decrease by at least 8% following treatment with the Hyper-CL™ lens only
* Corneal thickness decrease following treatment with the Hyper-CL™ lens only
* Measurement of distance visual acuity:

  o Best Corrected Distance Visual Acuity (BCDVA)
* Subject comfort

Subjects will be treated with:

A: Treatment with Hyper-CL™ lens only B: Treatment with Hyper-CL™ lens + salt solution C: Treatment with salt solution only Each subject will be treated with all three treatments according to his allocated regimen treatment.

1. Subject is over 18 years old
2. Subject with clinical corneal edema
3. Subject with visual acuity of 6/20 or worse (equivalent ETDRS)

1. Subject with active Herpes keratitis 2. Subject with scarred cornea 3. Subject who is suffering from erosions & infections of the cornea 4. Subject who require chronic administration of any topical ophthalmic beside lubrication eye drops and steroids or anti glaucoma drags 5. Subject who is currently participating or have participated in an investigational study, other than this study, within the past 60 days

Baseline: The visit will include subject's qualification assessment for inclusion/exclusion criteria as described above. Informed consent must be signed.

Complete anamnesis will be taken including subject's medical complaints, medical history, and medication use.

Ophthalmic examinations. Subject will be randomized to one of the 6 crossover regimen treatments.

Day 0: Subject will be asked to stop using any treatment for 7 days (beside steroid drops or anti glaucoma drops) and will have the following procedures/visits:

Day 7: subject will have clinical follow-up and will begin with first treatment (A, B or C) according to his treatment regimen.

Day 14: subject will have clinical follow-up and will stop the treatment. Day 21: subject will have clinical follow-up and will begin with the second treatment.

Day 28: subject will have clinical follow-up and will stop the treatment. Day 35: subject will have clinical follow-up and will begin the third treatment.

Day 42: subject will have clinical follow-up. All visits will include ophthalmic examinations, medications used and recording of adverse events. 42 days follow-up visit will include a satisfaction questionnaire.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is over 18 years old
2. Subject with clinical corneal edema
3. Subject with visual acuity of 6/20 or worse (equivalent ETDRS)

Exclusion Criteria:

1. Subject with active Herpes keratitis
2. Subject with scarred cornea
3. Subject who is suffering from erosions & infections of the cornea
4. Subject who require chronic administration of any topical ophthalmic beside lubrication eye drops and steroids or anti glaucoma drags
5. Subject who is currently participating or have participated in an investigational study, other than this study, within the past 60 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2013-07; Primary Completion 2014-01-31 (Actual); Study Completion 2014-04-30 (Actual)

PRIMARY OUTCOMES:
corneal thickness | 1 month
  Primary endpoint will be the percent of subjects with corneal thickness decrease of at least 8% during the one week treatment with the Hyper-CL™ lens + salt solution.

SECONDARY OUTCOMES:
visual acuity | 1 month
  Measurement of distance visual acuity:
  Best Corrected Distance Visual Acuity (BCDVA)

OTHER OUTCOMES:
Subject comfort | 1 month
  the comfort and pain relief

CONTACTS AND LOCATIONS:
Overall Officials: Irit Bachar, Md, Principal Investigator — Cornea physician
Locations (1):
- Rabin Medical Center, Petah Tikva, Israel